CLINICAL TRIAL: NCT06105281
Title: What Impact Does a Consultation With a Nurse Pain Specialist Have on Behaviour Towards Chronic Pain and Pain Intensity in Chronic Pain Patients?
Brief Title: Nurse Specialist Intervention Promoting Altered Coping and Treatment for Chronic Pain
Acronym: NURSIPACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Vitaz (Other)
Responsible Party: Principal Investigator, Filip Haegdorens, prof. dr. (PhD), Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NURSIPACT
Record Dates: First submitted 2023-10-12; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Monocentric Randomised controlled trail in the Vitaz Hospital of Sint-Niklaas. It will take place at the pain clinic where patient with chronic pain come for a treatment or infiltration against chronic pain. There will be two groups of patients, an intervention and an control arm with an equal allocation (1:1). The intervention and control arm will complete the study simultaneous. In each group will count 86 participance at the begin of the trail. This give us the possibility of 35% loss of follow up in each group, so that we can end the study with 64 participants in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The participants that only get the standard care in the pain clinic.
- The consultation with a pain specialist nurse (Experimental): When the participant receives a consultation with the pain specialist nurse ,there will be assessed if the patient knows what the procedure involves and what they can expect of it. To meet de expectations of the patient the nurse will explain the procedure and what they can expect. Further there will be an short education about what pain is and the physiology of chronic pain. Because chronic pain has a lot of influencing factors the nurse will explain the main factors.
  Interventions: Behavioral: The consultation with a pain specialist nurse

INTERVENTIONS:
Behavioral: The consultation with a pain specialist nurse — When the participant receives a consultation with the pain specialist nurse ,there will be assessed if the patient knows what the procedure involves and what they can expect of it. To meet de expectations of the patient the nurse will explain the procedure and what they can expect. Further there will be an short education about what pain is and the physiology of chronic pain. Because chronic pain has a lot of influencing factors the nurse will explain the main factors.
  Arms: The consultation with a pain specialist nurse

SUMMARY:
The aim of this study is to investigate of the implementation of an autonomous consultation with a nurse pain specialist for chronic pain patients has an influence on the behaviour towards the chronic pain. The trail will be done with patients that has planned an infiltration in a pain centre. Furthermore the pain intensity and patent satisfaction will be investigated as second outcomes.

During the consultation there will be explained what the patient can expect from the treatment in the pain clinic. What the patient expect from the infiltration will also be surveyed, so that it can be adjusted if necessary. In the end of the consultation there will be a brief explanation of chronic pain and the physiology as well als the different factors that have an influence on it.

This study is a monocentric randomised controlled trail of 172 participants, with an equal allocation (1:1). To collect the data there will be three different questionnaires for both groups. The first is a baseline measurement. The second will take place three weeks after the infiltration and the third ten weeks after the infiltration. This is in order to see if there is an evolution in the outcomes during time.

ELIGIBILITY:
Inclusion criteria:

* Patients that have an appointment for a treatment
* Patients with chronic pain, so 3 months or more and of functional dysfunction because of the pain.
* Patients that are receiving a spinal treatment form the cervical, thoracic or lumbar spine.
* The patient has to understand the Dutch language.

Exclusion criteria:

* Patients with a neurostimulator, an intrathecal medication pump or patients that already has an appointment at the consultation in the pain clinic. They have an doctor- patient relationship and that can cause bias.
* People who are legally incapable (persons younger then 18 years, persons with dementia, other cognitive diseases.
* People with facial pain. Here is the necessity of quick treatments. Or they already take place in other studies.
* People who are interned or detained. There is no possibility of follow-up.
* Palliative, oncologic or in hospital patients
* Patients who need a emergency treatment, because it is mostly acute or sub acute pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Behavior towards chronic pain | 7 months
  Pain solution questionaire (Pasol) by De Vlieger et al. (2006) - Min 0; Max 84 - Higher is better

CONTACTS AND LOCATIONS:
Overall Officials: Filip Haegdorens, PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Vitaz campus Sint-Niklaas, Sint-Niklaas, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No